CLINICAL TRIAL: NCT00891059
Title: The Role Of Cognitive Impairment In The Use Of The Diskus Inhaler
Acronym: Cognitive
Status: Completed | Type: Observational
Sponsor: Synergy Health Solutions (Other)
Responsible Party: Malcolm Fraser, MD, CMD, Synergy Health Solutions
Other Study IDs: DISKUS-01
Record Dates: First submitted 2009-04-27; First posted 2009-04-30 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Cognitive Impairment
Keywords: Cognitive Impairment; Diskus Inhaler; Nursing Home
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Placebo Diskus Inhaler

SUMMARY:
The Diskus Inhaler is administered by a nurse or medical technician in the Nursing Home (NH) setting. The administration of the medication from the Diskus Inhaler includes 4 steps: open, click, inhale, close. The only step that the resident must do is the "inhale" step, which includes holding one's breath for 10 seconds after the inhalation.

The investigators propose that properly trained and motivated nurses and medical technicians can successfully administer medication using the Advair Diskus to almost any mildly to moderately cognitively impaired resident who can follow the instruction- "inhale" and hold your breath for 10 seconds". The objective is to show that mild to moderate cognitive impairment should not be a barrier to the use of Diskus Inhaler. There will only be 1 consent visit and 1 evaluation visit per subject.

DETAILED DESCRIPTION:
Background and Objectives:

Approximately 1.6 million geriatric nursing home (NH) residents are living in about 17,000 Nursing Homes in the United States. This population (including those who live in Assisted Living Facilities [ALFs]) will increase significantly over the next 20 years as the "Baby Boomers" enter this age group. Associated with this will be an increasing number of cognitively impaired individuals with Chronic Obstructive Pulmonary Disease (COPD). As a nation, we will need to find effective and efficient means of caring for this growing population.

Sometimes there is an "intuitive anecdote"; a belief that mildly to moderately cognitively impaired individuals (score of 10 to 24 on the Mini Mental State Exam [MMSE]) are unable to synthesize and execute the instructions necessary for the successful use of the Diskus Inhaler for COPD. We propose a controlled assessment of DISKUS Inhaler use in mildly to moderately cognitively impaired residents living in NHs and ALFs.

The Diskus Inhaler is administered by a nurse or medical technician in the NH setting. The administration of the medication from the Diskus Inhaler includes 4 steps: open, click, inhale, close. The only step that the resident must do is the "inhale" step, which includes holding one's breath for 10 seconds after the inhalation.

We propose that properly trained and motivated nurses and medical technicians can successfully administer medication using the Advair Diskus to almost any mildly to moderately cognitively impaired resident who can follow the instruction- "inhale" and hold your breath for 10 seconds". The objective is to show that mild to moderate cognitive impairment should not be a barrier to the use of Diskus Inhaler.

Experimental Plan:

1. Equipment Diskus Inhalers filled with placebo only will be provided by GlaxoSmithKline.
2. Subjects:

   * Total number of subject will be 40
   * Subjects 18 and older will be selected from sites in the St. Petersburg, FL and Dayton, OH areas
   * No compensation will be given to subjects for participation
   * Subjects will spend about 15 -30 minutes at the one and only visit
   * The Mini Mental Status Exam (MMSE) will be administered to determine the degree of cognitive impairment
   * Subjects will be recruited by the investigators and study coordinators (SC) while visiting the NHs. No advertising will be done
3. Duration : Data collection will take 3 months with an additional 1 month data analysis period
4. Investigational Plan:

(i) There will be a Principal Investigator in each state - Dr Fraser in Florida and Dr Patel in Ohio. Fraser will also be the overall PI for the whole study.

(ii) Initial potential subjects will be drawn from the 2 practices that Dr Fraser and Dr Patel are part of. Initial screening will be based on informal chart review from the practices.

(iii) Initial contact of the potential subject/Legally Appointed Representative (LAR) will be from the PI/SubI/SC. The subject will be seen either in a Nursing Home (Bethany or Brooksville Health Care).

(iv) If the potential subject has a LAR, the LAR will be contacted first to obtain their informed consent before the study is discussed with the NH resident. The reason for this is that we do not want to appear to be pressuring the LAR to agree to the potential subject being enrolled. The reality is that living in a NH is monotonous and most NH patients enjoy doing something different. The LAR will be told that the patients' entering the study does not affect in any way the ongoing physician patient relationship

(v) If the LAR does not agree to allow the patient to be enrolled, the study will not be discussed with the patient, and if they ask why they can't do it, they will told that they are not eligible and they should discuss it with their LAR. They will NOT be told that the LAR had declined.

(vi) There will be 2 consents forms (Form A) ; one for the LAR and another version using simpler language (Assent - Form B) for all potential subjects to review and sign.

If the LAR agrees, once we have fulfilled the steps involving the LAR on the Informed Consent Form (ICF) Process and obtained written consent using Form A, then the study will be discussed with the potential subject and their assent will be requested using Assent Form B. If they do not want to participate, they will not be enrolled and they will not be regarded as enrolled until either we have obtained their assent by the completion of Assent Form B OR it is documented that they are unable to comprehend/sign Assent Form B

(vii) It is possible that since NHs/(Closed Congregate Retirement Centers)CCRCs are closed communities, word will get around and other NH residents, under the care of other physicians, will also want to be included. In this case, the PI/SubI/SC will ask the Nurses to obtain a written order from the attending physician, which will be placed on the patient's chart before the study is even discussed with the potential subject or the designated LAR.

(a) After the order is on the chart, the chart will be reviewed to determine if the patient is a potential subject. Then the stages d (iv) thru d (vi) will be followed.

(viii) After informed consent is obtained, the PI/Sub I/SC will meet the subject and review the chart in order to confirm eligibility.

1. The resident will be asked to take a deep breath and hold it while the PI/Sub I/SC counts to 10.
2. If the subject is able to hold their breath for 10 seconds, then the subject will be given the MMSE.
3. If the score on the MMSE falls between 10 and 24 inclusively, the subject will be instructed on the use of the Diskus Inhaler.
4. The PI/Sub I/SC will demonstrate the open, click, inhale, and close phases and then ask the resident to repeat the actions.
5. The PI/Sub I/SC may repeat the demonstration 2 more times, (for a total of 3 demonstrations) if necessary, for the resident to complete all 4 tasks successfully.
6. The PI/SubI/SC will allow 1-2 minutes between each attempt if the resident is showing signs of shortness of breath. The PI/Sub I/SC will then rate each step on the Diskus Inhaler Evaluation Scale (Appendix I).
7. The rating will end after the resident successfully completes all 4 phases or the resident 3 unsuccessfully attempts, whichever comes first.
8. The rater will then complete a global assessment of the use of the Diskus Inhaler, indicating overall whether the subject adequately or inadequately used the Diskus Inhaler
9. The subject will be told that they have completed the study and thanked for their cooperation. They will be asked if they have any questions and all questions will be answered before the PI/SubI/SC leaves the room
10. The unit charge nurse will be told that the resident has completed the study and thanked

(xii) The LARs/potential subjects will be told that there is no financial benefit to either of them in any way and that the study will take a maximum of 30 mins. They will be told that there is no other direct benefit of any type to them but the knowledge gained may help companies design delivery mechanisms which other cognitively impaired people, like the subject, may benefit from in the future.

(xii). There are no other study requirements.

e. Chronology of Study: (i) A total of 40 subjects will be studied - 20 in Florida and 20 in Ohio. If for any reason the sites in either state are unable to enroll 20, then the sites in the other state will make up the deficiency.

The following timeline is anticipated after receiving IRB approval:

Week 1-4: Print forms, team meetings by phone between the 2 sites to review protocol and ensure uniformity.

Week 5-12: Enroll subjects and perform study

Week13-18: Perform statistical analysis, prepare and submit final report.

(ii) Number of visits. Screening/ Consent explained 1 Consent obtained/ Evaluation visit 1

There will be a minimum of 3 days between the 2 visits.

f. Power Analysis:

We determined the sample size if the 2 groups differ by as little as 50%. The estimated sample size for two-sample comparison of proportions:

Test Ho: p1 = p2, where p1 is the proportion in population 1 and p2 is the proportion in population 2

Assumptions:

alpha = 0.0500 (two-sided) power = 0.9000 p1 = 1.0000 p2 = 0.5000 n2/n1 = 1.00

Estimated required sample sizes:

n1 = 18 n2 = 18

We expect to say that we examined for differences in Diskus use between groups that could be as small as 50% with confidence (P<.05 in two-tail testing & with a Power of 0.90).

g. Safety Monitoring:

Since there is no intervention, there will be no safety monitoring. Adverse events (AEs) will not be recorded. Serious adverse events (SAEs) will be captured only if the PI or Sub-I feels the event is related to the study procedures.

h. Confidentiality protection:

All data will be identified with the resident's initials and a 4 digit subject number. No names will be used. The data will be kept with the PI/Sub I/SC and brought back from the NH to the research facility and stored in a locked area. No one other than study staff will have access to the data collected. All data will be collected on paper; no electronic files will be used.

Risk Analysis/Informed Consent:

Since a placebo will be inhaled for a maximum of 3 times, we believe there to be no risk to the residents.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women residing in a NH or ALF
* Mini Mental Status Exam (MMSE) score between 10 and 24 inclusive
* Able to hold breath for at least 10 seconds
* Able to speak and understand English

Exclusion Criteria:

* Current or history of Diskus use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nursing Home Residents with Mini Mental Status Exam (MMSE) score between 10 and 24 inclusive with convenience sampling or invitation to volunteer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The objective is to show that mild to moderate cognitive impairment should not be a barrier to the use of Diskus Inhaler. | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm R Fraser, MD, Principal Investigator — President, Synergy Health Solutions
Locations (2):
- United States (2):
  - Brooksville Health Care Center, Brooksville, Florida
  - Bethany Village, Centerville, Ohio